CLINICAL TRIAL: NCT00361725
Title: Comparative Study of the Protein C Pathway in Septic and Non Septic Patients
Brief Title: Comparative Study of the Protein C Pathway in Septic and Non Septic Patients With Organ Failure
Status: Terminated | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Other Study IDs: PROCAS
Record Dates: First submitted 2006-08-07; First posted 2006-08-08 (Estimated); Last update posted 2006-08-15 (Estimated); Status verified 2006-06

CONDITIONS: Severe Sepsis; Organ Failure
Keywords: severe sepsis; organ failure; activated protein C; thrombomodulin; EPCR
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
This is a comparative study performed in 3 groups of patients/subjects: 30 severe sepsis patients, 30 non-septic patients with organ failure, 30 healthy subjects.

The only intervention is a venous blood sampling at the onset of the disease.

The purpose of the study is to compare the PC pathway and expression and inflammatory genes between the 3 groups. The main hypothesis is that systemic inflammatory response and exacerbated coagulation activation are non specific of an infection as a triggering event.

DETAILED DESCRIPTION:
analysis of the PC pathway

* PC activity
* PS activity
* soluble thrombomodulin
* soluble EPCR
* activated protein C
* quantitative flow cytometry on monocytes (thrombomodulin and EPCR)
* whole blood mRNA (Tissue factor, thrombomodulin and EPCR)
* inflammatory gene expression analysis by MLPA

ELIGIBILITY:
Inclusion Criteria:

* severe sepsis patients or:
* non-septic acute organ failure patients or:
* healthy subjects matched for age and sex with severe sepsis patients

Exclusion Criteria:

* criteria for organ failure lasting for more than 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2003-03; Study Completion 2003-10

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc DIEHL, MD, Principal Investigator — Assistance Publique Hopitaux de Paris

REFERENCES:
- [Result] Borgel D, Clauser S, Bornstain C, Bieche I, Bissery A, Remones V, Fagon JY, Aiach M, Diehl JL. Elevated growth-arrest-specific protein 6 plasma levels in patients with severe sepsis. Crit Care Med. 2006 Jan;34(1):219-22. doi: 10.1097/01.ccm.0000195014.56254.8a. PMID 16374177
- [Derived] Borgel D, Bornstain C, Reitsma PH, Lerolle N, Gandrille S, Dali-Ali F, Esmon CT, Fagon JY, Aiach M, Diehl JL. A comparative study of the protein C pathway in septic and nonseptic patients with organ failure. Am J Respir Crit Care Med. 2007 Nov 1;176(9):878-85. doi: 10.1164/rccm.200611-1692OC. Epub 2007 Aug 2. PMID 17673691